CLINICAL TRIAL: NCT00558545
Title: A Phase 1-2, Multicenter, Open-Label Study of the X-Linked Inhibitor of Apoptosis (XIAP) Antisense AEG35156 Given in Combination With Weekly Paclitaxel in Patients With Advanced Breast Cancer
Brief Title: A Phase 1-2, XIAP Antisense AEG35156 With Weekly Paclitaxel in Patients With Advanced Breast Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Avastin approved for first-in-line treatment.
Sponsor: Aegera Therapeutics (Industry)
Responsible Party: Jacques Jolivet, VP Clinical, Aegera Therapeutics Inc.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEG35156-202
Record Dates: First submitted 2007-11-13; First posted 2007-11-15 (Estimated); Last update posted 2009-12-02 (Estimated); Status verified 2009-11

CONDITIONS: Human Mammary Carcinoma
Keywords: Breast; paclitaxel; antisense; oligonucleotide
MeSH Terms: conditions — Breast Neoplasms | interventions — AEG 35156

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: AEG35156 — AEG35156 will be given as a 2-hour intravenous infusion once weekly only on weeks when paclitaxel is administered, with a 2-hour loading dose given daily in the 2 days immediately prior to Day 1 (on Days -2 and -1) only in Cycle 1.

SUMMARY:
This is an open-label multicenter, phase 1-2 study. Following determination of the recommended AEG35156 dose in combination with weekly paclitaxel in the initial Phase 1 part of this study, additional patients will be enrolled in the Phase 2 part of the study to assess the activity of the combination in advanced breast cancer.

DETAILED DESCRIPTION:
Breast cancer is the most common cancer in women in the United States, the second most common cause of cancer death, and the main cause of death in women ages 45 to 55. In 2006, 212,920 American women will be diagnosed with breast cancer, and 40,970 will die from this disease.[1]. Fewer than 10 percent of women present with metastatic disease at the time of diagnosis. However, the majority of women who relapse after initial definitive therapy for early stage or locally advanced disease will do so with disseminated metastatic disease rather than an isolated local recurrence. Treatment for metastatic disease is palliative in intent and will usually involve hormone therapy and/or chemotherapy with or without trastuzumab. Active chemotherapy agents include anthracyclines, taxanes, vinorelbine, alkylating agents and antimetabolites. Taxanes have become the cornerstone of first-line treatment for metastatic breast cancer. Weekly doses of paclitaxel can be administered continuously for several weeks with a remarkable lack of myelosuppression [2]. Weekly paclitaxel (80 mg/m2) was directly compared to every three-week therapy (175 mg/m2) in 585 women with metastatic breast cancer. Weekly therapy was associated with a significantly higher response rate (40 versus 28 percent) and longer TTP (nine versus five months), but similar overall survival and worse neurotoxicity [3]. Since patients with metastatic breast cancer are unlikely to be cured of their disease [4], they should be considered candidates for a clinical trial.

ELIGIBILITY:
Inclusion Criteria:

* Patients with histologically or cytologically confirmed breast adenocarcinoma who are candidates for paclitaxel single agent chemotherapy for metastatic breast cancer
* ECOG performance < 2
* One or more metastatic tumors measurable by RECIST criteria on CT scan or MRI (Phase 2 part only)
* Life expectancy of at least 6 months
* Age > 18 years
* Signed, written IRB-approved informed consent
* A negative serum pregnancy test (if applicable)
* Acceptable liver function:
* Bilirubin within normal limit
* AST (SGOT), ALT (SGPT) and Alkaline phosphatase < 2.0 times the institution's upper limit of normal
* Acceptable renal function:
* Serum creatinine within normal limits, OR calculated creatinine clearance > 60 mL/min/1.73 m2 for patients with creatinine levels above institutional normal
* Acceptable hematologic status:
* Granulocyte > 1500 cells/uL
* Platelet count > 100,000 plt/uL
* Hemoglobin > 9.0 g/dL
* Acceptable coagulation status:
* PT within normal limits
* PTT within normal limits
* For women of child-bearing potential, the use of effective contraceptive methods during the study
* Prior radiotherapy is allowed provided disease progression outside the radiation field has been documented, and treatment completed at least 2 weeks prior to registration

Exclusion Criteria:

* Prior taxane chemotherapy for metastatic disease.
* More than one prior chemotherapy regimen for metastatic disease
* Active progressive brain metastases including the presence of any related symptoms or need for corticosteroids. A CT or MRI scan of the head is necessary in patients with a history of brain metastases to document the stability of prior lesions
* Grade > 2 peripheral neuropathy
* Known bleeding diathesis or concurrent treatment with anticoagulants except patients on non-therapeutic line maintenance coumadin
* Pregnant or nursing women. NOTE: Women of child-bearing potential must agree to use adequate contraception (sterile or surgically sterile; hormonal or barrier method of birth control; or abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Active, uncontrolled bacterial, viral, or fungal infections, requiring systemic therapy
* Known infection with HIV, hepatitis B, or hepatitis C
* Serious nonmalignant disease that could compromise protocol objectives in the opinion of the investigator and/or the sponsor
* Patients who are currently receiving any other investigational agent. Subjects who have used a previous antisense oligonucleotide in the last 90 days will be excluded
* Unwillingness or inability to comply with procedures required in this protocol
* Any deviation from these inclusion/exclusion criteria must be discussed with the sponsor prior to enrolling patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Estimated)
Dates: Start 2007-11; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
To determine the recommended dose of AEG35156 when used in combination with weekly paclitaxel and at the dose enhance the clinical benefit rate (CBR) of paclitaxel in patients with advanced breast cancer. | 2 years

SECONDARY OUTCOMES:
To determine progression-free survival. | 2 years
To establish the pharmacokinetics of AEG35156 and paclitaxel when used in combination. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: David M Loesch, MD, Principal Investigator — Central Indiana Cancer Centers; Jacques Jolivet, MD, FACP, Study Director — Aegera Therapeutics, Inc.
Locations (10):
- United States (10):
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Cancer Centers of Florida, P.A., Ocoee, Florida
  - Central Indiana Cancer Center, Indianapolis, Indiana
  - New York Oncology & Hematology P. C., Albany Cancer Center, Albany, New York
  - Dayton Oncology & Hematology, P.A., Dayton, Ohio
  - Cancer Centers of the Carolinas, Greenville, South Carolina
  - Sammons Cancer Center, Dallas, Texas
  - Tyler Cancer Center, Tyler, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, P. C., Vancouver, Washington

REFERENCES:
- [Background] Jemal A, Siegel R, Ward E, Murray T, Xu J, Smigal C, Thun MJ. Cancer statistics, 2006. CA Cancer J Clin. 2006 Mar-Apr;56(2):106-30. doi: 10.3322/canjclin.56.2.106. PMID 16514137
- [Background] Perez EA, Vogel CL, Irwin DH, Kirshner JJ, Patel R. Multicenter phase II trial of weekly paclitaxel in women with metastatic breast cancer. J Clin Oncol. 2001 Nov 15;19(22):4216-23. doi: 10.1200/JCO.2001.19.22.4216. PMID 11709565
- [Background] Seidman, A., et al., CALGB 9840: Phase III study of weekly paclitaxel via 1-hour infusion versus standard 3h infusion every third week in the treatment of metastatic breast cancer (MBC), with trastuzumab (T) for HER2 positive MBC and randomized for T in HER2 normal MBC. Proc Am Soc Clin Oncol, 2004. 23: p. 6s.
- [Background] Greenberg PA, Hortobagyi GN, Smith TL, Ziegler LD, Frye DK, Buzdar AU. Long-term follow-up of patients with complete remission following combination chemotherapy for metastatic breast cancer. J Clin Oncol. 1996 Aug;14(8):2197-205. doi: 10.1200/JCO.1996.14.8.2197. PMID 8708708